CLINICAL TRIAL: NCT02977533
Title: A Randomized, Double-blind, Placebo-controlled Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Subcutaneous Dose of GZ402668 in Men and Women With Progressive Multiple Sclerosis
Brief Title: A Single Ascending Dose Study of GZ402668 in Patients With Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDU14981; 2016-002415-18 (EudraCT Number); U1111-1184-8607 (Other: UTN)
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GZ402668 (Experimental): Dose 1 (up to a maximum optional Dose 2) will be given as a single subcutaneous administration under fed conditions. Acyclovir will be given twice daily starting on Day 1 and continuing for 28 days after investigational medicinal product administration.
  Interventions: Drug: GZ402668; Drug: Acyclovir
- Placebo (Placebo Comparator): A dose of matching placebo will be given as a single subcutaneous administration under fed conditions. Acyclovir will be given twice daily starting on Day 1 and continuing for 28 days after investigational medicinal product administration.
  Interventions: Drug: Placebo; Drug: Acyclovir

INTERVENTIONS:
Drug: GZ402668 — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: GZ402668
Drug: Placebo — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Placebo
Drug: Acyclovir — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To assess the safety and tolerability of GZ402668 after a single subcutaneous (SC) dose in men and women with progressive multiple sclerosis.

Secondary Objectives:

To assess in men and women with progressive multiple sclerosis:

* The pharmacokinetic (PK) parameters of GZ402668 after a single SC dose.
* The pharmacodynamic (PD) response to GZ402668 after a single SC dose.

DETAILED DESCRIPTION:
The total study duration from screening for a patient can be approximately up to 8 weeks. Upon completion of this trial, patients treated with GZ402668 will be required to enroll in a 4 year safety follow-up study for continued safety observation.

ELIGIBILITY:
Inclusion criteria :

* Male or female adult with a diagnosis of progressive multiple sclerosis (MS) including primary progressive MS, secondary progressive MS, or progressive relapsing MS.
* Aged between 18 and 65 years, inclusive.
* Body weight greater than 40.0 kg.
* Female patients of child bearing potential must use 2 highly effective contraception methods.
* Male patients, whose partners are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, 2 highly effective contraception methods. Males patient, whose partners are pregnant, must use, during sexual intercourse, a condom from the inclusion up to 4 months after investigational medicinal product administration.
* Males patient who has agreed not to donate sperm for 4 months after product administration.

Exclusion criteria:

* Significant medical diseases or conditions, including poorly controlled hypertension, cardiovascular disease, inflammatory disorders, immunodeficiency, autoimmune disease, renal failure, liver dysfunction, cancer (except treated basal skin cell carcinoma), or active infection.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day.
* If female, pregnancy, lactating, or breast-feeding.
* Patients with relapsing-remitting MS.
* Treatment with natalizumab, methotrexate, azathioprine, or cyclosporine in the past 6 months.
* Treatment with mitoxantrone, cyclophosphamide, cladribine, rituximab or any other immunosuppressant or cytotoxic therapy (other than steroids) in the last 12 months, or determined by the treating physician to have residual immune suppression from these treatments.
* Treatment with glatiramer acetate or interferon beta in the past 4 weeks.
* Treatment with fingolimod within the past 2 months.
* Treatment with dimethyl fumarate in past 4 weeks.
* Treatment with teriflunomide within the past 12 months unless patient has completed an accelerated clearance with cholestyramine.
* Previous treatment with alemtuzumab.
* Live, attenuated vaccine within 3 months prior to the randomization visit, such as varicella-zoster, oral polio, and rubella vaccines.
* Clinically significant abnormality in thyroid function.
* Inability to undergo magnetic resonance imaging with gadolinium administration.
* Hypersensitivity or contraindication to acyclovir.
* Known bleeding disorder.
* Significant autoimmune disease.
* Active infection or at high risk for infection.
* Latent or active tuberculosis.
* Major psychiatric disorder that is not adequately controlled by treatment.
* Epileptic seizures that are not adequately controlled by treatment.
* Prior history of invasive fungal infections.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events | 4 weeks

SECONDARY OUTCOMES:
Assessment of PK parameter: maximum concentration (Cmax) | 4 weeks
Assessment of PK parameter: area under curve (AUC) | 4 weeks
Number of participants with lymphocyte depletion | 4 weeks
Number of participants with anti-drug antibodies | 4 weeks
Number of participants with injection site reactions | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Albach FN, Geier C, Keicher C, Posch MG, Schreiber SJ, Grutz G, Akyuz L, Luo X, Le-Halpere A, Truffinet P, Wagner F. Phase 1 Trials of Gatralimab, a Next-Generation Humanized Anti-CD52 Monoclonal Antibody, in Participants with Progressive Multiple Sclerosis. Neurol Ther. 2024 Dec;13(6):1607-1625. doi: 10.1007/s40120-024-00659-w. Epub 2024 Sep 9. PMID 39251561